CLINICAL TRIAL: NCT03545269
Title: A Multi-Center, Active-Controlled, Open-Label, Phase Ⅱ Trial to Compare the Efficacy and Safety for Treatment of Autologous Chondrocytes Implantation With CartiLife Versus Microfracture for Patient With Chondral Defects in the Knee
Brief Title: Study to Assess the Efficacy and Safety of Treatment of Articular Cartilage Lesions With CartiLife®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosolution Co., Ltd. (Industry)
Collaborators: Kyunghee University Medical Center (Other); Gangnam Severance Hospital (Other); Severance Hospital (Other); Ewha Womans University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCTT-CTL-021
Record Dates: First submitted 2018-03-08; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Articular Cartilage Lesion of the Knee
Keywords: Degenerative Arthritis; Autologous Chondrocyte Implantation; Cartilage defects; Cartilage lesion; Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Intervention Model Description: Biological: CartiLife® Procedure: CartiLife® is beads (1.0 to 1.5 mm in diameter) in suspension, developed from autologous chondrocytes. The beads are implanted in a volume of 1 cm3 per the capacity of the syringe to the affected area through injection along with a fibrin adhesive through minimal arthrotomy.
  Active comparator: Microfracture The surgery is performed by arthroscopy, after the joint is cleaned of calcified cartilage. Through use of an awl, the surgeon creates tiny fractures in the subchondral bone plate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CartiLife® (Experimental)
  Interventions: Drug: CartiLife®
- Microfracture (Active Comparator)
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Drug: CartiLife® — CartiLife® is beads (1.0 to 1.5 mm in diameter) in suspension, developed from autologous chondrocytes. The beads are implanted the volume of 1 cm3 per the capacity of the syringe to the affected area through injection with fibrin adhesive through minimal arthrotomy.
  Arms: CartiLife®
Procedure: Microfracture — The surgery is performed by arthroscopy, after the joint is cleaned of calcified cartilage. Through use of an awl, the surgeon creates tiny fractures in the subchondral bone plate.
  Arms: Microfracture

SUMMARY:
The purpose of this study is to assess the safety and efficacy of implanting bead-type autologous chondrocyte (CartiLife®) obtained by culturing expanded costal chondrocytes of the patient with a chondral defect in the knee. The patients will be assessed clinically using MRI, clinical, biochemical and International Knee Documentation Committee(IKDC) outcomes preoperatively as well as 8, 24 and 48 weeks postoperatively to assess the relief of symptoms and joint function.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged between 19 and 65
* Defect size: 2 to 10 ㎠ on the unilateral knee cartilage (up to 4 ㎤ in volume)
* Defect: isolated International Cartilage Repair Society(ICRS) Grade III or IV single defect chondral lesion on articular cartilage
* The joint space is maintained over 50% relative to baseline
* Patients that are able to walk without aid
* Patients that agree to abide by strict rehabilitation protocols and follow-up programs
* Patients who provide written consent to the participation of the clinical trial

Exclusion Criteria:

* Patients with inflammatory articular diseases such as rheumatoid arthritis or gouty arthritis
* Kellgren and Lawrence grade ≥ 3
* Patients with arthritis associated with autoimmune diseases
* Patients hypersensitive to bovine protein
* Patients with Haemophilia or markedly reduced immune function
* Patients hypersensitive to antibiotics like gentamicin
* Patients with arterial bleeding and severe venous bleeding
* Patients with other diseases including tumors except for cartilaginous defects of joints
* Patients with a history of radiation treatment and chemotherapy within the past two years
* Patients who are pregnant, nursing a baby or likely to get pregnant
* Patients who participate in concurrent clinical trials or previous clinical trials within 30 days of administration
* Other cases where the investigator deems the patient ineligible for participation

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue) | Baseline to 48 weeks
  Changes in MOCART scores during each visit

SECONDARY OUTCOMES:
Lysholm Score | Baseline to 48 weeks
  Changes in Lysholm Scores during each visit
IKDC (International Knee Documentation Committee Score) | Baseline to 48 weeks
  Changes in IKDC scores during each visit
KOOS (Knee injury Osteoarthritis Outcome Score) | Baseline to 48 weeks
  Changes in KOOS during each visit
VAS (100 mm Pain Visual Analogue Scale) | Baseline to 48 weeks
  Changes in VAS during each visit
ROM (Range Of Motion) | Baseline to 48 weeks
  Changes in ROM during each visit
Adverse events | Baseline to 48 weeks
  Number of adverse events
X-ray | Baseline to 48 weeks
  Changes in structure during each visit

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Ho, MD, PhD, Principal Investigator — Kyunghee University Medical Center; Jong Hyeok Choi, MD, PhD, Principal Investigator — Severance Hospital; Jae-Doo Yoo, MD, PhD, Principal Investigator — Ewha Womans University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoon KH, Lee J, Park JY. Costal Chondrocyte-Derived Pellet-Type Autologous Chondrocyte Implantation Versus Microfracture for the Treatment of Articular Cartilage Defects: A 5-Year Follow-up of a Prospective Randomized Trial. Am J Sports Med. 2024 Feb;52(2):362-367. doi: 10.1177/03635465231222797. Epub 2024 Jan 17. PMID 38230875
- [Derived] Yoon KH, Yoo JD, Choi CH, Lee J, Lee JY, Kim SG, Park JY. Costal Chondrocyte-Derived Pellet-Type Autologous Chondrocyte Implantation versus Microfracture for Repair of Articular Cartilage Defects: A Prospective Randomized Trial. Cartilage. 2021 Dec;13(1_suppl):1092S-1104S. doi: 10.1177/1947603520921448. Epub 2020 Jun 1. PMID 32476445